CLINICAL TRIAL: NCT00101283
Title: Pemetrexed Plus Gemcitabine Or Carboplatin In Patients With Advanced Malignant Mesothelioma: A Randomized Phase II Trial
Brief Title: Pemetrexed Plus Gemcitabine or Carboplatin for Patients With Advanced Malignant Pleural Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); North Central Cancer Treatment Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000401795; U10CA021115 (NIH); E1B03 (Other: ECOG); E1B03 (Other: NCCTG)
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Results first posted 2010-03-04 (Estimated); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Mesothelioma
Keywords: advanced malignant mesothelioma; recurrent malignant mesothelioma
MeSH Terms: conditions — Mesothelioma; Mesothelioma, Malignant | interventions — Pemetrexed; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pemetrexed/Carboplatin (Experimental): Pemetrexed disodium 500 mg/m2 IV over 10 minutes and carboplatin to area under the curve (AUC) 5 IV over 30 minutes on day 1 of a 21-day cycle.
  Interventions: Drug: pemetrexed disodium; Drug: carboplatin
- Pemetrexed/Gemcitabine (Experimental): Pemetrexed disodium 500 mg/m2 IV over 10 minutes on day 1 and gemcitabine 1000 mg/m2 IV over 30 minutes on days 1 and 8 of a 21-day cycle.
  Interventions: Drug: pemetrexed disodium; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: pemetrexed disodium — 500 mg/m2 IV over 10 minutes on day 1 of a 21-day cycle
  Other Names: Alimta; MTA; LY231514
Drug: gemcitabine hydrochloride — 1000 mg/m2 IV over 30 minutes on days 1 and 8 of a 21-day cycle
  Other Names: Gemzar
  Arms: Pemetrexed/Gemcitabine
Drug: carboplatin — Given by IV over 30 minutes at an area under the curve (AUC) of 5 on day 1 of a 21-day cycle
  Other Names: CBDCA; Paraplatin; JM-8; NSC-241240
  Arms: Pemetrexed/Carboplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as pemetrexed disodium, gemcitabine, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. It is not yet known whether giving pemetrexed disodium with gemcitabine is more effective than giving pemetrexed disodium with carboplatin in treating malignant pleural mesothelioma.

PURPOSE: This randomized phase II trial is studying pemetrexed disodium with gemcitabine and pemetrexed disodium with carboplatin to see how well the combinations work compared to historical controls in treating patients with advanced malignant pleural mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the response rates in patients with advanced malignant mesothelioma of the pleura treated with pemetrexed disodium combined with either gemcitabine or carboplatin.

Secondary

* Assess the toxic effects of these regimens in these patients.
* Estimate survival time in patients treated with these regimens.
* Correlate smoking status with outcome in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms. While randomized, the study is not a comparative study. Rather, outcomes on each arm will be compared to a historical control rate from previous studies. Randomization allows simultaneous testing of two experimental arms.

* Arm I: Patients receive intravenous (IV) pemetrexed disodium over 10 minutes and carboplatin IV over 30 minutes on day 1.
* Arm II: Patients receive pemetrexed disodium as in arm I and gemcitabine IV over 30 minutes on days 1 and 8.

In both arms, treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Beginning approximately 5-10 days before the start of chemotherapy and continuing until approximately 3 weeks after completion of chemotherapy, all patients receive oral folic acid once daily and cyanocobalamin (vitamin B12) intramuscularly every 9 weeks.

Patients are followed every 3 months for 2 years and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 32-60 patients (16-30 per treatment arm) will be accrued for this study within 12.8-27.0 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced mesothelioma of the pleura
* Measurable disease, as defined by RECIST criteria, within 4 weeks of randomization. Patients with pleural rinds not measurable by RECIST were eligible if disease was evaluable within 4 weeks of randomization using mesothelioma response criteria
* May have undergone pleurodesis. If pleurodesis was performed, there must have been at least a 2-week delay before Pemetrexed administration. A CT must have been performed after 2 weeks after pleurodesis to serve as the baseline scan.
* ECOG Performance Status of 0 or 1
* Normal organ and marrow function, as defined by:

  * Absolute neutrophil count ≥ 1,500/ul
  * Platelet count ≥ 100,000/ul
  * Bilirubin ≤ 1.5 times upper limit of normal (ULN)
  * AST and ALT ≤ 3 times ULN (5 times ULN if liver has tumor involvement)
  * Albumin ≥ 2.5 g/dL
  * Creatinine clearance ≥ 45 mL/min or Creatinine ≤ 2.0 g/dL
* Age 18 years and over
* Able to take folic acid and cyanocobalamin (vitamin B12)
* Willing and able to take dexamethasone
* Women of childbearing potential and sexually active men were required to use contraception during and for the first 3 months after the study

Exclusion Criteria

* A candidate for curative surgery
* Prior radiation therapy to the target lesion, unless the lesion was clearly progressing per RECIST criteria after prior radiation and the interval between the most recent radiation therapy and enrollment was at least 4 weeks
* Prior systemic chemotherapy for mesothelioma. Prior intracavitary cytotoxic drugs or immunomodulators were not permitted, unless given for the purpose of pleurodesis.
* Active infection or serious concomitant systemic disorder
* Second primary malignancy, other than in situ malignancies or adequately treated basal cell carcinoma of the skin or other malignancy treated at least 3 years previously with no evidence of recurrence.
* Treatment with an investigational agent within 4 weeks before enrollment
* Known or suspected brain metastases
* Women must not be pregnant or breastfeeding
* Obviously malnourished or with a weight loss of greater than 10% in the preceding 6 weeks
* Aspirin or other nonsteroidal anti-inflammatory drugs for 2 days before, during, and for 2 days after each administration of pemetrexed disodium (5 days before, during, and 2 days after each administration of pemetrexed disodium for piroxicam, naproxen, diflunisal, or nabumetone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-02-23 (Actual); Primary Completion 2009-09 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasser H. Hanna, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center; Scott Okuno, MD, Study Chair — Mayo Clinic
Locations (115):
- United States (115):
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on November 1, 2005, accrued its first patient on February 23, 2006, suspended to accrual on July 12, 2007 for response evaluation, and closed to accrual on April 1, 2008.
Groups:
- Pemetrexed/Carboplatin: Pemetrexed disodium 500 mg/m2 IV over 10 minutes and carboplatin to AUC 5 IV over 30 minutes on day 1 of a 21-day cycle.
Period: Overall Study
Arm/Group | Pemetrexed/Carboplatin | Pemetrexed/Gemcitabine
Started | 16 | 16
Began Treatment | 16 | 13
Completed | 16 | 13
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Insurance Refusal | 0 | 1
Not completed — Prostate Cancer Recurrence | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemetrexed/Carboplatin | Pemetrexed/Gemcitabine | Total
Number analyzed (Participants) | 16 | 13 | 29
Age, Continuous [Median (Full Range); unit: years] | 72 [55 to 78] | 68 [53 to 80] | 71 [53 to 80]
Sex: Female, Male [Count of Participants; unit: Participants] — Gender of participants who began treatment.
  Participants
    Female | 2 | 12 | 14
    Male | 14 | 1 | 15

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response by RECIST Criteria (Version 1.0)
Description: Number of eligible, treated participants in each response category by RECIST criteria. Response categories represent best response for each patient prior to progression.
Time Frame: Assessed every 2 cycles (6 weeks) while on treatment, then every 3 months for 2 years, then every 6 months for 1 year until disease progression
Population: The population consisted of all eligible, treated patients. 3 patients randomized to pemetrexed/gemcitabine who withdrew prior to treatment are excluded.
Measure: Number; unit: eligible, treated participants
Arm/Group | Pemetrexed/Carboplatin | Pemetrexed/Gemcitabine
Number analyzed (Participants) | 16 | 13
eligible, treated participants
  Partial Response | 3 | 0
  Stable Disease | 7 | 6
  Progression | 5 | 5
  Unevaluable | 1 | 2
Statistical Analysis 1: Comparison: Pemetrexed/Carboplatin; The treatment was to be considered promising if a true response rate of 40% or higher was observed, whereas a rate of 15% or less would not be of interest. 3 or more responses were required to expand accrual to a second stage. This expansion did not occur; Test type: Superiority or Other; Overall Response Percent = 18.8, 90% CI 2-sided [5.4 to 41.7] — Overall response percent for Pemetrexed/Carboplatin arm (percent of eligible, treated patients with complete or partial response)
Statistical Analysis 2: Comparison: Pemetrexed/Gemcitabine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Overall Response Percent = 0.0, 90% CI 2-sided [0.0 to 20.6] — Overall response percent for Pemetrexed/Gemcitabine arm (percent of eligible, treated patients with complete or partial response)

2. Secondary Outcome: Overall Survival
Description: Time from randomization to death. Patients alive at last follow-up were censored.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 1 year
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed/Carboplatin | Pemetrexed/Gemcitabine
Number analyzed (Participants) | 16 | 13
Months | 13.0 [5.6 to 21.9] | 6.0 [3.9 to 14.0]

3. Secondary Outcome: Progression-Free Survival
Description: Time from randomization to the earlier of disease progression or death. Patients alive and progression-free at last follow-up were censored.
Time Frame: Assessed every 3 months for 2 years, then every 6 months for 1 year
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed/Carboplatin | Pemetrexed/Gemcitabine
Number analyzed (Participants) | 16 | 13
Months | 4.1 [1.7 to 6.6] | 3.3 [1.6 to 5.2]

ADVERSE EVENTS:
Time Frame: Assessed every cycle (21 days) while on treatment and for 30 days after the end of treatment.
Arm/Group | Pemetrexed/Carboplatin | Pemetrexed/Gemcitabine
Serious Adverse Events (participants affected / at risk) | 10/16 | 13/13
Other Adverse Events (participants affected / at risk) | 16/16 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed/Carboplatin (N=16) | Pemetrexed/Gemcitabine (N=13)
Anemia (Blood and lymphatic system disorders) | 3 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 10
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2
Fatigue (General disorders) | 2 | 3
Anorexia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Elevated bilirubin (Investigations) | 1 | 0
Arachnoiditis/meningismus/radiculitis (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Chest/thoracic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed/Carboplatin (N=16) | Pemetrexed/Gemcitabine (N=13)
Allergic rhinitis (Immune system disorders) | 1 | 0
Hearing loss (without baseline audiogram, not in monitoring program) (Ear and labyrinth disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 14 | 12
Hemolysis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 13 | 11
Lymphopenia (Blood and lymphatic system disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 11 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 7
Fatigue (General disorders) | 15 | 12
Fever w/o neutropenia (General disorders) | 3 | 3
Insomnia (General disorders) | 1 | 3
Rigors/chills (General disorders) | 2 | 1
Sweating (General disorders) | 1 | 1
Weight gain (General disorders) | 1 | 1
Weight loss (General disorders) | 3 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritis/itching (Skin and subcutaneous tissue disorders) | 2 | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5 | 5
Skin - other (Skin and subcutaneous tissue disorders) | 1 | 1
Hot flashes (Endocrine disorders) | 1 | 0
Anorexia (Gastrointestinal disorders) | 5 | 9
Constipation (Gastrointestinal disorders) | 6 | 5
Dehydration (Gastrointestinal disorders) | 0 | 2
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 3 | 2
Distention/bloating, abdominal (Gastrointestinal disorders) | 0 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0
Muco/stomatitis (symptom), oral cavity (Gastrointestinal disorders) | 0 | 1
Muco/stomatitis (symptom), pharynx (Gastrointestinal disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 9 | 4
Taste disturbance (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 3 | 4
GI - other (Gastrointestinal disorders) | 0 | 1
Colitis, infectious (Gastrointestinal disorders) | 1 | 0
Infection w/ gr 0-2 neutrophils, sinus (Infections and infestations) | 2 | 0
Edema, limb (Blood and lymphatic system disorders) | 0 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 11
Elevated alkaline phosphatase (Metabolism and nutrition disorders) | 3 | 9
Elevated ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 5 | 6
Elevated AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 3 | 6
Elevated bilirubin (Metabolism and nutrition disorders) | 1 | 2
Elevated creatinine (Investigations) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 2
Hemoglobinuria (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal/soft tissue - other (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 2
Depression (Nervous system disorders) | 0 | 1
Neuropathy, sensory (Nervous system disorders) | 1 | 1
Tearing (Eye disorders) | 1 | 0
Ocular - other (Eye disorders) | 1 | 0
Abdomen, pain (Gastrointestinal disorders) | 1 | 0
Bone, pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest/thoracic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Extremity - limb, pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint, pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Liver, pain (Hepatobiliary disorders) | 0 | 1
Muscle, pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 1
Vascular - other (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No